CLINICAL TRIAL: NCT01321138
Title: Comparison of Incidence of Femoral Neuropathy After Anterior Cruciate Ligament Reconstruction With Femoral Nerve Block Versus Patient-controlled Analgesia (PCA)
Brief Title: Femoral Neuropathy After Anterior Cruciate Ligament Reconstruction: Femoral Nerve Block vs Patient-controlled Analgesia (PCA)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, Eric Albrecht, Chef de Clinique, Centre Hospitalier Universitaire Vaudois
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: CHUV-75-10
Record Dates: First submitted 2011-03-22; First posted 2011-03-23 (Estimated); Last update posted 2015-11-30 (Estimated); Status verified 2015-11

CONDITIONS: Femoral Neuropathy
Keywords: Electrophysiological study; Nerve block; Analgesia, Patient-Controlled; Anterior cruciate ligament
MeSH Terms: conditions — Femoral Neuropathy; Agnosia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Femoral nerve block (Active Comparator): Continuous femoral nerve block with bolus of ropivacaine 0.5% and then continuous infusion of ropivacaine 0.2 % 4 - 6 ml/h, associated with paracetamol and ibuprofen. Each group will contain 30 patients.
  Interventions: Procedure: Femoral nerve block
- PCA morphine (Placebo Comparator): Patients with iv morphine with self administration with a PCA-system, associated with paracetamol and ibuprofen.
  Interventions: Procedure: PCA morphine

INTERVENTIONS:
Procedure: Femoral nerve block — The femoral nerve block will be performed with ultrasound 30 minutes before the intervention
  Other Names: ANY
  Arms: Femoral nerve block
Procedure: PCA morphine — Postoperative analgesia with self-administration iv morphine
  Other Names: ANY
  Arms: PCA morphine

SUMMARY:
Femoral neuropathy after anterior cruciate ligament reconstruction with femoral nerve block may be as high as 24% at 6 postoperative weeks when evaluated prospectively and systematically through a clinical neurological and an electroneuromyography (ENMG). It is still unclear whether this neuropathy is the result of the surgery, especially the Tourniquet, or the block nerve. The goal of this study is to define the etiology of this postoperative neuropathy.

DETAILED DESCRIPTION:
Anterior cruciate ligament reconstruction is associated with moderate to severe postoperative pain. Among different analgesic strategies, continuous femoral nerve block is reported as an efficient method, reducing opioid consumption and allowing rapid rehabilitation; however, patients may develop a transient neuropathy after surgery, which could have a significant impact on active patients, particularly on athletes who need immediate rehabilitation and who will put their knee to greater use during the postoperative period. This study is designed to compare the incidence of femoral neuropathy in two groups of patients: one with a femoral nerve block, and one with a PCA of morphine (self-iv administration of morphine). All patients will have a clinical neurological exam with a preoperative ENMG in order to rule out a pre-existing neuropathy. Another clinical neurological exam with ENMG will be performed between 4 and 6 weeks and, if pathological, repeated at 6 months, 9 months and 12 months. The operation will be done under general anesthesia for all patients.

ELIGIBILITY:
Inclusion Criteria:

* patients planned for anterior cruciate ligament reconstruction
* ASA 1 and 2
* age 16 years and more

Exclusion Criteria:

* peripheral neuropathy
* pre-existing femoral neuropathy
* diabetes mellitus
* alcoholism
* drug addiction
* cancer with chemotherapy
* chronic pain state

Ages: 16 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 74 (Actual)
Dates: Start 2011-04; Primary Completion 2014-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Incidence of femoral neuropathy | 6 weeks
  Clinical neurological exam (diminished or absent patellar reflex, or sensory loss in the femoral nerve territory) and ENMG (Axon loss ratio, Hofmann reflex, coumpound muscle action potentials, any fibrillation potentials of the muscle at rest) at 6 postoperative weeks. A control will be done at 3 months if a neuropathy is present.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Albrecht, MD, Principal Investigator — Department of Anesthesia, Centre Hospitalier Universitaire Vaudois and University of Lausanne
Locations (1):
- Centre Hospitalier Universitaire Vaudois and University of Lausanne, Lausanne, Canton of Vaud, Switzerland

REFERENCES:
- [Derived] Stebler K, Martin R, Kirkham KR, Kuntzer T, Bathory I, Albrecht E. Electrophysiological Study of Femoral Nerve Function After a Continuous Femoral Nerve Block for Anterior Cruciate Ligament Reconstruction: A Randomized, Controlled Single-Blind Trial. Am J Sports Med. 2017 Mar;45(3):578-583. doi: 10.1177/0363546516669715. Epub 2016 Nov 13. PMID 27836905